CLINICAL TRIAL: NCT04713696
Title: Using Functional Movement Patterns to Investigate the Impact of Core Stability on Hitting Mechanics and Bat Swing Velocity in High School Baseball Players
Brief Title: Core Stability for Baseball Batting in Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Yi Liang Kuo, Assistant Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B-ER-108-072
Record Dates: First submitted 2021-01-03; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Athletes; Adolescent
Keywords: Batting mechanics; Bat-swing velocity; Baseball; Lumbopelvic control; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional training (Experimental): Participants received functional training
  Interventions: Other: Functional training
- Routine training (Active Comparator): Participants received routine training
  Interventions: Other: Routine training

INTERVENTIONS:
Other: Functional training — Functional training refers to exercises that targets the muscles of the lumbopelvic-hip complex in order for them to more appropriately support and control the spine.
  Arms: Functional training
Other: Routine training — Routine training refers to general exercises that perform before and after practice, including jogging, stretching and strengthening exercises for upper and lower extremities
  Arms: Routine training

SUMMARY:
Baseball batting is important to winning the games. Baseball batting is achieved by proximal-to-distal sequencing of body movements and controlled by the neuromuscular system. Poor lumbopelvic control could influence production and transfer of energy in the kinetic chain. This study aims to investigate the effects of functional movement training on hitting mechanics and bat swing velocity in high school baseball players.

ELIGIBILITY:
Inclusion Criteria:

* Sport specialization in baseball batting
* Active players on baseball teams

Exclusion Criteria:

* History of surgery in the lumbar area
* Severe musculoskeletal or neurological symptoms that interfere with participation in competition, training or tests

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-12 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Bat-swing velocity | Changes from baseline to 8 weeks post intervention
  Maximal bat swing velocity during baseball batting measured by the VICON motion analysis system
Batting movement | Changes from baseline to 8 weeks post intervention
  Batting movement measured by the VICON motion analysis system

SECONDARY OUTCOMES:
Dynamic balance | Changes from baseline to 8 weeks post intervention
  Dynamic balance measured by the Y-balance Test (YBT)
Functional performance | Changes from baseline to 8 weeks post intervention
  Functional performance measured by Functional Movement Screen (FMS)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Liang Kuo, PT, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University, Tainan, Taiwan